CLINICAL TRIAL: NCT03529786
Title: A Retrospective and Cross-sectional Study to Evaluate Neurodevelopmental Status in Pediatric Subjects With Severe Mucopolysaccharidosis Type II (Hunter Syndrome)
Brief Title: Mucopolysaccharidosis Type II Natural History
Status: Completed | Type: Observational
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-121-002
Record Dates: First submitted 2018-02-13; First posted 2018-05-18 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Mucopolysaccharidosis II
Keywords: Hunter Syndrome; Natural History; Iduronate-2-sulfatase; glycosaminoglycans
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective: An observational medical records review study (data collected retrospectively) in subjects with the severe form of MPS II.

SUMMARY:
Mucopolysaccharidosis type II (MPS II), also known as Hunter syndrome, is caused by a deficiency of iduronate-2-sulfatase (IDS) leading to an accumulation of glycosaminoglycans (GAGs) in tissues of MPS II patients, resulting in characteristic storage lesions and diverse disease sequelae, and in patients with the more severe form of the disease, irreversible neurocognitive decline and higher morbidity and mortality than in patients with the attenuated form of the disease.

There is currently limited information on the natural history of MPS II, especially with respect to neurocognitive decline in patients with the more severe form of the disease. This study is planned to be an observational medical records review study (data collected retrospectively and no investigational product treatment or procedures) in subjects with the severe form of MPS II. Collectively, the data may inform the design of future MPS II gene therapy treatment studies and may be utilized as historical comparative control data.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of MPS II confirmed by enzyme activity as measured in plasma, fibroblasts, or leukocytes
2. The subject has at least one of the neurocognitive assessments listed below, which occurred prior to age 6 and in or after 2006 in their medical records.

   1. Bayley Scales of Infant and Toddler Development (BSID), any version
   2. Differential Ability Scale (DAS), any version
   3. Griffiths Mental Development Scale (GMDS), any version
   4. Kaufman Assessment Battery for Children (KABC), any version
   5. Kinder Infant Development Scale (KIDS)
   6. Kyoto Scale of Psychological Development (KSPD), any version
   7. Leiter International Performance Scale (LIPS), any version
   8. Mullen Scales of Early Learning (MSEL), any version
   9. Vineland Adaptive Behavior Scales (VABS), any version
   10. Wechsler Intelligence Scale for Children (WISC), any version
   11. Wechsler Preschool and Primary Scale of Intelligence (WPPSI), any version
3. If the subject has undergone hematopoietic stem cell transplantation (HSCT), they must have at least one neurocognitive assessment prior to HSCT.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children diagnosed with Mucopolysaccharidosis type II (MPS II), also known as Hunter syndrome
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Cognitive function over time, as indicated by results of neurocognitive measures documented in medical chart. | Up to 10 years old
  There are 10 neurocognitive measures that provide intelligence quotients (IQ) scores and/or developmental quotients (DQ) scores.

SECONDARY OUTCOMES:
Prevalence of general organ involvement and specific characteristics of severe MPS II as documented in medical chart. | Up to 10 years old
  Documentation in medical chart regarding date and age of onset of:
  Disease Characteristics, General Appearance, Neurologic/Psychiatric, Cardiovascular, Ocular, Musculoskeletal, Auditory, Respiratory, Gastroenterology/Urinary, Interventional Medications, Other Interventions, ER and Hospitalization History, MRI History, ECG History
Age of onset of general organ involvement and specific characteristics of severe MPS II as documented in medical chart. | Up to 10 years old
  Documentation in medical chart regarding date and age of onset of:
  Disease Characteristics, General Appearance, Neurologic/Psychiatric, Cardiovascular, Ocular, Musculoskeletal, Auditory, Respiratory, Gastroenterology/Urinary, Interventional Medications, Other Interventions, ER and Hospitalization History, MRI History, ECG History

CONTACTS AND LOCATIONS:
Locations (3):
- Children's Hospital of Pittsburgh - UPMC: Program for Neurodevelopment in Rare Disorders, Pittsburgh, Pennsylvania, United States
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Manchester Centre for Genomic Medicine, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided